CLINICAL TRIAL: NCT00675285
Title: Effects of Oral Montelukast on Airway Inflammation in Children With Mild Asthma
Brief Title: Effects of Montelukast in Children With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Paolo Montuschi, M.D. Associate Professor of Pharmacology, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A/1064/2004; NCT00496496 (obsolete NCT alias)
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Asthma
Keywords: airway inflammation; childhood asthma; fractional exhaled nitric oxide; leukotriene receptor antagonists; lung function
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: montelukast sodium
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: montelukast sodium — one tablet 5 mg once/day for 4 weeks
  Arms: 1
Drug: placebo — one tablet 5 mg once/day for 4 weeks
  Arms: 2

SUMMARY:
Leukotriene receptor antagonists (LTRAs) reduce fractional exhaled nitric oxide (FENO) concentrations in children with asthma, but the effect of LTRA withdrawal on FENO and lung function is unknown. We will aim to study the effect of treatment and withdrawal of montelukast, a LTRA, on airway inflammation as reflected by FENO and lung function in children with asthma.

A double-blind, randomized, placebo controlled, parallel group study will be undertaken in 18 atopic children with mild persistent asthma who will be treated with oral montelukast (5 mg/day for 4 weeks) and 18 atopic children with mild persistent asthma who will receive matching placebo.

A follow-up visit will be performed 2 weeks after montelukast or placebo withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Children 6 to 14 yrs old, step 1 and step 2 GINA (Global INitiative for Asthma) guidelines
* exhaled nitric oxide (NO) >20 PPB at visit 2
* symptoms more often than twice a day, FEV1 equal or higher than 80% of predicted value and reversibility equal or higher than 12% to salbutamol, or a positive provocation test with methacholine, or exercise
* no regular medication, inhaled short-acting beta-2 agonists for symptom relief

Exclusion Criteria:

* Patient is hospitalized
* Patient has FEV1 < 80% predicted on visit 1
* Patient has 2 or more nighttime awakenings for asthma per week or pef variability 30% or more
* upper respiratory infection in the previous 3 weeks
* treatment with glucocorticoids or LTRAs in the previous 4 weeks
* treatment with inhaled glucocorticoids for more than 4 weeks in the previous year

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2005-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
post-treatment fractional exhaled nitric oxide

SECONDARY OUTCOMES:
fractional exhaled nitric oxide 2 weeks after montelukast withdrawal
post-treatment FEV1
post-treatment FVC
post-treatment FEV1/FVC
post-treatment FEF25%-75%
FEV1 2 weeks after montelukast withdrawal
FVC 2 weeks after montelukast withdrawal
FEV1/FVC 2 weeks after montelukast withdrawal
FEF25%-75% 2 weeks after montelukast withdrawal
asthma exacerbation rate

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Montuschi, M.D., Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Catholic University of the Sacred Heart, Rome, Italy